CLINICAL TRIAL: NCT02031302
Title: RESPOND: Re-positionable Lotus Valve System - Post Market Evaluation of Real World Clinical Outcomes
Brief Title: RESPOND Post Market Study
Acronym: RESPOND
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TP6461
Record Dates: First submitted 2014-01-06; First posted 2014-01-09 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Aortic Valve Stenosis
Keywords: Lotus; Valve; Real world; Aortic stenosis; High risk
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lotus Valve: All subjects who are candidates for Transcatheter Aortic Valve Implantation (TAVI), signed the Informed Consent Form (ICF) and are selected to receive a Lotus Valve.
  Interventions: Device: Lotus Valve System
- Lotus with Depth Guard: All subjects who are candidates for Transcatheter Aortic Valve Implantation (TAVI), signed the Informed Consent Form (ICF) and are selected to receive a Lotus with Depth Guard.
  Interventions: Device: Lotus Valve System

INTERVENTIONS:
Device: Lotus Valve System — The Lotus Valve System is indicated to improve aortic valve function for symptomatic subjects with severe calcific aortic stenosis (aortic valve area [AVA] of <1.0 cm2 or index of <0.6 cm2/m2) who are at high risk for standard surgical valve replacement.

SUMMARY:
The purpose of the RESPOND post market study is to collect real world clinical and device performance outcomes data with the Lotus Valve System used in routine clinical practice to demonstrate that the commercially available Lotus Valve System is a safe and effective treatment for patients with severe calcific aortic stenosis.

DETAILED DESCRIPTION:
The RESPOND study is a prospective, open label, single arm, multi-center, observational post market study designed to collect real world clinical and device performance outcomes data of the commercially available Lotus Valve used in routine clinical practice for the treatment of severe calcific aortic stenosis. Approximately 1000 real-world, consecutive subjects will be enrolled at up to 50 study centers in Europe, Asia Pacific and Central/South America.

All enrolled subjects will be contacted for follow-up at 30 days, 1, 2, 3, 4 and 5 years post index valve implantation. Follow-up visit at 1 year post valve implantation should be conducted via outpatient clinic visit. Follow-up visits at 30 days and 2 through 5 years may be conducted in person (preferred) and via telephone interview. Subjects who are not implanted with a Lotus Valve will be followed for safety through 30 days after the initial attempted index procedure.

Collection of safety events will include any serious adverse event (SAE) that led to death, serious adverse device effect (SADE), adverse device effect (ADE), unanticipated serious adverse device effect (USADE), and all Valve Academic Research Consortium (VARC) events regardless of seriousness and device relationship through 5 year follow-up.

The RESPOND study will be conducted in accordance with the International Organization for Standardization (ISO) 14155: 2011; ethical principles that have their origins in the Declaration of Helsinki; the relevant parts of the International Conference on Harmonization (ICH) Guidelines for Good Clinical Practices (GCP); and pertinent individual country/state/local laws and regulations.

An additional cohort of approximately 50 subjects will be enrolled at up to 6 study centers in Europe after enrollment in the main cohort is completed to assess center-driven implantation technique with the commercially available Lotus Valve with Depth Guard technology.

ELIGIBILITY:
Subjects will be evaluated for eligibility by the clinical center's heart team per the local standard of practice in accordance with the Directions for Use.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects who are candidates for Transcatheter Aortic Valve Implantation (TAVI), signed the Informed Consent Form (ICF) and are selected to receive a Lotus Valve will be evaluated for enrollment in this study.
Sampling Method: Probability Sample
Enrollment: 1064 (Actual)
Dates: Start 2014-05-27 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Van Mieghem, MD, Principal Investigator — Erasmus Medical Center; Volkmar Falk, MD, PhD, Principal Investigator — German Heart Center Berlin
Locations (41):
- Colombia (2):
  - Angiografia de Occidente S.A., Cali
  - Fundacion Cardiovascular de Colombia, Floridablanca
- Finland (2):
  - Helsinki University Central Hospital/Meilahti Hospital, Helsinki
  - Turku University Hospital, Turku
- Germany (14):
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Krankenhaus d. Barmherzigen Brüder, Trier, Rhineland-Palatinate
  - Herz-Kreislauf-Zentrum Segeberger Kliniken GmbH, Bad Segeberg
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Charité Campus Virchow Klinikum, Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - Herz- und Gefäß-Klinik Bonn, Bonn
  - Asklepios Klinik St. Georg, Hamburg
  - Herzzentrum Universitat Leipzig, Leipzig
  - Deutsches Herzzentrum München, Munich
  - University Hospital Munich, Munich
  - Universitätsklinikum Rostock, Rostock
  - HELIOS Clinic, Siegburg
  - Universitätsklinikum Ulm, Ulm
- Rabin Medical Center, Petah Tikva, Israel
- Italy (4):
  - IRCC Policlinico San Donato, Milan, Mi
  - Azienda Ospedaliera Universtitaria di Padova, Padua, PD
  - Azienda Ospedaliera Universtiatia Pisana (AOUP) Ospedale Cisanello, Pisa, PI
  - Ospedale San Raffaele, Milan
- Netherlands (2):
  - Dept. of Cardiology Sint-Antonius ziekenhuis, Nieuwegein, EM
  - Erasmus Medical Center, Rotterdam
- Waikato Hospital, Hamilton, New Zealand
- Haukeland universitetssjukehus, Bergen, Norway
- Poland (2):
  - I Klinika Kardiologii Uniwersytetu Medycznego W Poznaiu, Poznan
  - National Institute of Cardiology, Warsaw
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Policlinica Gipuzkoa, San Sebastián
- Sahlgrenska University Hospital, Gothenburg, Sweden
- INSELSPITAL - Universitätsspital Bern, Bern, Switzerland
- United Kingdom (8):
  - John Radcliffe Infirmary Oxford II, Oxford, England
  - Royal Sussex County Hospital, Brighton
  - Leeds Teaching Hospitals NHS, Leeds
  - Glenfield Hospital, Leicester
  - Clinical Trials Practitioner, London
  - King's College Hospital London, London
  - Cardiovascular & Cell Sciences Research Institute, London
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html).

REFERENCES:
- [Derived] Van Mieghem NM, Wohrle J, Hildick-Smith D, Bleiziffer S, Blackman DJ, Abdel-Wahab M, Gerckens U, Linke A, Ince H, Wenaweser P, Allocco DJ, Meredith IT, Falk V. Use of a Repositionable and Fully Retrievable Aortic Valve in Routine Clinical Practice: The RESPOND Study and RESPOND Extension Cohort. JACC Cardiovasc Interv. 2019 Jan 14;12(1):38-49. doi: 10.1016/j.jcin.2018.10.052. PMID 30621976
- [Derived] Falk V, Wohrle J, Hildick-Smith D, Bleiziffer S, Blackman DJ, Abdel-Wahab M, Gerckens U, Linke A, Ince H, Wenaweser P, Allocco DJ, Dawkins KD, Van Mieghem NM. Safety and efficacy of a repositionable and fully retrievable aortic valve used in routine clinical practice: the RESPOND Study. Eur Heart J. 2017 Dec 1;38(45):3359-3366. doi: 10.1093/eurheartj/ehx297. PMID 28651336

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 1014 subjects enrolled at 41 centers in Germany, UK, Italy, Colombia, Finland, The Netherlands, Poland, Spain, Israel, New Zealand, Norway, Sweden and Switzerland between 27 May 2014 and 01 Feb 2016.
  50 subjects were enrolled in the cohort with the Lotus Depth Guard valve between 13 Jun 2016 and 31 Oct 2016.
Pre-assignment Details: Lotus Valve cohort: 1 subject had the 1 year visit on 25SEP2015, but died on 02OCT2015, that's why the disposition table only shows 115 subjects died prior to 1 year Follow-up performed . A total of 116 subjects died through 1 year (365 days) post procedure (as treated population). 120 of 1002 patients died according to the ITT population.
Groups:
- Lotus Valve: All subjects who are candidates for Transcatheter Aortic Valve Implantation (TAVI), signed the Informed Consent Form (ICF) and are selected to receive a Lotus Valve.
  Lotus Valve System: The Lotus Valve System is indicated to improve aortic valve function for symptomatic subjects with severe calcific aortic stenosis (aortic valve area [AVA] of <1.0 cm2 or index of <0.6 cm2/m2) who are at high risk for standard surgical valve replacement.
  These are the 1 year outcome.
- Lotus With Depth Guard: All subjects who are candidates for Transcatheter Aortic Valve Implantation (TAVI), signed the Informed Consent Form (ICF) and are selected to receive a Lotus with Depth Guard.
  Lotus Valve System: The Lotus Valve System is indicated to improve aortic valve function for symptomatic subjects with severe calcific aortic stenosis (aortic valve area [AVA] of <1.0 cm2 or index of <0.6 cm2/m2) who are at high risk for standard surgical valve replacement.
  These are the 30 days outcome. Study ended at 30 days. No 1 year data collected.
Period: Overall Study
Arm/Group | Lotus Valve | Lotus With Depth Guard
Started | 1014 | 50
Completed | 850 | 50
Not Completed | 164 | 0
Not completed — Death | 115 | 0
Not completed — Not treated with study valve system | 18 | 0
Not completed — Missed Follow Up | 27 | 0
Not completed — Lost to Follow-up | 4 | 0

BASELINE CHARACTERISTICS:
Population: This is a post-market trial. Only 996 out of 1014 subjects are treated with the Lotus valve in the Lotus Valve arm (as treated population). In the Lotus with Depth Guard arm all 50 subjects are treated with the device.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lotus Valve | Lotus With Depth Guard | Total
Number analyzed (Participants) | 996 | 50 | 1046
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.8 (6.5) | 80.9 (8.2) | 80.8 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 506 | 23 | 529
  Male | 490 | 27 | 517
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
European System for Cardiac Operative Risk Evaluation (EuroSCORE 2011) [Mean (Standard Deviation); unit: units on a scale] — The European System for Cardiac Operative Risk Evaluation is a risk model where if a risk factor is present in a subject, a weight or number is assigned. The weights are added to give an approximate percent predicted mortality. A higher score means a higher risk and a lower score means a lower risk.
  units on a scale | 8.0 (8.4) | 3.3 (1.7) | 7.8 (8.2)
New York Heart Association (NYHA) Classification [Number; unit: participants] — New York Heart Association Classification is a system for defining cardiac disease and related functional limitations into four broad categorizations. The categories range from NYHA I (No limitations) to NYHA IV (inability to carry out any physical activity without discomfort).
  participants
    NYHA I | 34 | 1 | 35
    NYHA II | 248 | 22 | 270
    NYHA III | 577 | 25 | 602
    NYHA IV | 66 | 1 | 67
    Not done | 71 | 1 | 72
Society of Thoracic Surgeons (STS) Risk Score [Mean (Standard Deviation); unit: units on a scale] — The Society of Thoracic Surgeons Score is a risk model used to predict a subject's risk of mortality and morbidities for the most commonly performed cardiac surgeries. The model is a percentage score from 0 to 100 where a lower score means a lower risk and higher score means a higher risk.
  units on a scale | 6.0 (6.9) | 4.4 (3.1) | 5.9 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: The primary endpoint is all-cause mortality at 30 days after the implant procedure. The primary safety endpoint will be evaluated on an intention-to-treat (ITT) basis (all subjects enrolled, whether or not a Lotus Valve is implanted). All-cause mortality at 30 days after the implant procedure will be compared to a pre-specified performance goal.
Time Frame: 30 Days
Population: The primary endpoint analysis is based on the ITT population (1014) through 30 days; 9 subjects out of 1014 subjects are excluded from the analysis because they don't have sufficient follow up, their last follow up days are less than 23 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotus Valve | Lotus With Depth Guard
Number analyzed (Participants) | 1005 | 50
Participants | 26 | 0
Statistical Analysis 1: Comparison: Lotus Valve; Note: the 95% CI is from Clopper-Pearson Exact Method. The analysis was only done for the Lotus valve arm as the Lotus with Depth Guard arm has not sufficient power for this statistical analysis; Test type: Other — One-sided Clopper-Pearson 98.699% upper bound; p < .0001, Chi-squared — The proportion of patients who experience an event through 30 days post-procedure out of the patients who have either had an event within 30 days post-procedure or who were event-free with last follow-up at least 23 days post-procedure; One-sided Clopper-Pearson 98.699% upper bound: 4.11% Performance goal is 14%

2. Primary Outcome: All-cause Mortality
Description: The primary endpoint is all-cause mortality at 1 year after the implant procedure. The primary safety endpoint will be evaluated on an intention-to-treat (ITT) basis (all subjects enrolled, whether or not a Lotus Valve is implanted).
  A total of 116 subjects died through 1 year (365 days) post procedure (as treated population). 4 additional patients died but were not treated with the study valve system (ITT population).
  The Lotus Valve cohort is an ongoing study in it's 4 year follow up. The Lotus with Depth Guard cohort ended after 30 day follow up, therefore we have no data at 1 year.
Time Frame: 1 Year
Population: The primary endpoint analysis is based on the ITT population (1014) through 1 year; 12 subjects out of 1014 subjects are excluded from the analysis because they don't have sufficient follow up, their last follow up days are less than 320 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotus Valve
Number analyzed (Participants) | 1002
Participants | 120

3. Secondary Outcome: Percentage of Participants With Events Included in the Safety Composite Endpoint of All-Cause Mortality and Disabling Stroke
Description: All subjects who are candidates for transcatheter aortic valve implantation (TAVI), signed the Informed Consent Form (ICF) and are selected to receive a Lotus Valve will be evaluated for enrollment in this study (as treated population) The Lotus Valve cohort is an ongoing study in it's 4 year follow up. The Lotus with Depth Guard cohort ended after 30 day follow up, therefore we have no data at 1 year.
Time Frame: 30 Days and 1 year
Population: The Safety composite of all-cause mortality and disabling stroke analysis is based on the as treated population for the Lotus valve arm (996) through 1 year; 8 subjects out of 996 subjects are excluded from the analysis because they don't have sufficient follow up; their last follow up days are less than 320 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotus Valve | Lotus With Depth Guard
Number analyzed (Participants) | 988 | 50
Participants
  30 day outcome | 41 | 1
  1 year outcome: number analyzed (Participants) | 988 | 0
  1 year outcome | 135 | 0

4. Secondary Outcome: In-hospital Mortality
Description: In-hospital mortality till discharge
Time Frame: Duration of hospital stay, an expected average of 2 days
Population: The In-hospital till discharge analysis is based on the as treated population for the Lotus valve arm (996). In the Lotus with Depth Guard arm are all patients treated with the device.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotus Valve | Lotus With Depth Guard
Number analyzed (Participants) | 996 | 50
Participants | 18 | 0

5. Secondary Outcome: Percentage of Participants With Events Included in the VARC Efficacy Composite Endpoint
Description: The VARC efficacy composite at 1 year, including all-cause mortality; all stroke (disabling and non-disabling); re-hospitalization for valve-related symptoms or worsening congestive heart failure (NYHA class III or IV); and prosthetic valve-related dysfunction (mean aortic valve gradient ≥20 mmHg, effective orifice area (EOA) ≤0.9-1.1 cm2 and/or Doppler velocity index (DVI) <0.35 m/s, AND/OR moderate or severe prosthetic valve aortic regurgitation)
Time Frame: 1 Year
Population: The Lotus Valve cohort is an ongoing study in it's 4 year follow up. The Lotus with Depth Guard cohort ended after 30 day follow up, therefore we have no data at 1 year. 443 patients had no Echo analysis and therefore no data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotus Valve
Number analyzed (Participants) | 553
Participants | 200

6. Secondary Outcome: Patients With Valve Safety Composite Outcomes at 1 Year
Description: Time related valve safety composite outcomes at 1 year, including structural valve deterioration (valve-related dysfunction requiring repeat procedure [TAVI or SAVR]); prosthetic valve endocarditis; prosthetic valve thrombosis; thromboembolic events (e.g. stroke) and VARC bleeding, unless clearly unrelated to valve therapy based on investigator assessment (e.g. trauma).
  The Lotus Valve cohort is an ongoing study in it's 4 year follow up. The Lotus with Depth Guard cohort ended after 30 day follow up, therefore we have no data at 1 year.
Time Frame: 1 Year
Population: The analysis of patients with valve safety composite outcomes at 1 year is based on the as treated population for the Lotus valve arm (996) through 1 year; 8 subjects out of 996 subjects are excluded from the analysis because they don't have sufficient follow up; their last follow up days are less than 320 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotus Valve
Number analyzed (Participants) | 988
Participants | 219

7. Secondary Outcome: Patients With VARC Safety Composite Outcomes at 30 Days
Description: Patients with VARC safety composite outcomes at 30 days. VARC safety composite endpoints are defined as:
  * Life-threatening bleeding
  * Acute kidney injury-Stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure (BAV, TAVI, or SAVR)
  * New conduction disturbances (LBBB, AVB, RBBB) and need for permanent pacemaker implantation
Time Frame: 30 Days
Population: The analysis of patients with valve safety composite outcomes at 30 days based on the as treated population for the Lotus valve arm (996) through 30 days. In the Lotus with Depth Guard arm are all patients treated with the device.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotus Valve | Lotus With Depth Guard
Number analyzed (Participants) | 996 | 50
Participants | 334 | 10

8. Secondary Outcome: Patients With Moderate and Severe Paravalvular Aortic Valve Regurgitation
Description: Grade of paravalvular aortic valve regurgitation pre-discharge as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory. The moderate and severe paravalvular aortic regurgitation rate will be compared to a pre-specified performance goal.
  We don't have a powered analysis for the PVL for RESPOND study.
Time Frame: Duration of hospital stay, an expected average of 2 days
Population: 62 patients had no data available for the analysis in the Lotus Valve arm. 13 patients had no data for the analysis in the Lotus with Depth Guard arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotus Valve | Lotus With Depth Guard
Number analyzed (Participants) | 934 | 37
Participants | 179 | 13

ADVERSE EVENTS:
Time Frame: 1 year for the LOTUS valve group. The Lotus Depth guard group was only assessed up to 30 days.
Description: Lotus Valve cohort: 1 subject had the 1 year visit on 25SEP2015, but died on 02OCT2015, that's why the disposition table only shows 115 subjects died prior to 1 year Follow-up performed . A total of 116 subjects died through 1 year (365 days) post procedure (as treated population). 120 of 1002 patients died according to the ITT population.
Groups:
- Lotus Valve (30 Day Follow Up); Lotus Valve (1 Year Follow Up): All subjects who are candidates for Transcatheter Aortic Valve Implantation (TAVI), signed the Informed Consent Form (ICF) and are selected to receive a Lotus Valve.
  Lotus Valve System: The Lotus Valve System is indicated to improve aortic valve function for symptomatic subjects with severe calcific aortic stenosis (aortic valve area [AVA] of <1.0 cm2 or index of <0.6 cm2/m2) who are at high risk for standard surgical valve replacement.
- Lotus With Depth Guard (30 Day Follow Up): All subjects who are candidates for Transcatheter Aortic Valve Implantation (TAVI), signed the Informed Consent Form (ICF) and are selected to receive a Lotus with Depth Guard.
  Lotus Valve System: The Lotus Valve System is indicated to improve aortic valve function for symptomatic subjects with severe calcific aortic stenosis (aortic valve area [AVA] of <1.0 cm2 or index of <0.6 cm2/m2) who are at high risk for standard surgical valve replacement.
Arm/Group | Lotus Valve (30 Day Follow Up) | Lotus Valve (1 Year Follow Up) | Lotus With Depth Guard (30 Day Follow Up)
All-Cause Mortality (participants affected / at risk) | 22/987 | 116/988 | 0/50
Serious Adverse Events (participants affected / at risk) | 426/1014 | 525/1014 | 14/50
Other Adverse Events (participants affected / at risk) | 96/1014 | 99/1014 | 7/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lotus Valve (30 Day Follow Up) (N=1014) | Lotus Valve (1 Year Follow Up) (N=1014) | Lotus With Depth Guard (30 Day Follow Up) (N=50)
Total (Cardiac disorders) | 327 (354) | 382 (451) | 9 (9)
Atrioventricular block complete (Cardiac disorders) | 149 (149) | 155 (155) | 6 (6)
Conduction disorder (Cardiac disorders) | 57 (57) | 58 (58) | 1 (1)
Cardiac failure (Cardiac disorders) | 7 (7) | 46 (47) | 0 (0)
Bundle branch block left (Cardiac disorders) | 19 (19) | 24 (24) | 0 (0)
Atrioventricular block (Cardiac disorders) | 20 (20) | 20 (20) | 1 (1)
Bradycardia (Cardiac disorders) | 12 (12) | 14 (14) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 12 (12) | 13 (13) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 11 (12) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 11 (11) | 11 (11) | 0 (0)
Pericardial effusion (Cardiac disorders) | 10 (10) | 11 (11) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 9 (9) | 9 (9) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 7 (7) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 6 (6) | 7 (7) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 7 (7) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 5 (5) | 5 (5) | 0 (0)
Cardiac arrest (Cardiac disorders) | 6 (6) | 5 (5) | 0 (0)
Trifascicular block (Cardiac disorders) | 4 (4) | 4 (4) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Aortic valve disease (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Cardiac asthma (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Electromechanical dissociation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular asystole (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Total (Injury, poisoning and procedural complications) | 50 (52) | 66 (70) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 25 (26) | 29 (30) | 2 (2)
Vascular procedure complication (Injury, poisoning and procedural complications) | 9 (9) | 11 (11) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 7 (7) | 8 (8) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Renal injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Total (Nervous system disorders) | 34 (35) | 56 (63) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 17 (17) | 30 (32) | 2 (2)
Cerebral infarction (Nervous system disorders) | 5 (5) | 6 (6) | 1 (1)
Hemiparesis (Nervous system disorders) | 5 (5) | 5 (5) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Total (General disorders) | 27 (27) | 54 (54) | 1 (1)
Death (General disorders) | 1 (1) | 19 (19) | 0 (0)
Catheter site haemorrhage (General disorders) | 14 (14) | 14 (14) | 1 (1)
Multi-organ failure (General disorders) | 3 (3) | 8 (8) | 0 (0)
Catheter site haematoma (General disorders) | 6 (6) | 7 (7) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site haematoma (General disorders) | 1 (1) | 1 (1) | 0 (0)
Obstruction (General disorders) | 1 (1) | 1 (1) | 0 (0)
Puncture site haemorrhage (General disorders) | 1 (1) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Total (Infections and infestations) | 5 (5) | 32 (33) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 10 (10) | 0 (0)
Endocarditis (Infections and infestations) | 2 (2) | 8 (8) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 6 (6) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cardiac valve abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Total (Vascular disorders) | 32 (34) | 30 (33) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 7 (7) | 7 (7) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 4 (4) | 4 (4) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 4 (4) | 4 (4) | 0 (0)
Femoral artery dissection (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 3 (3) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)
Aneurysm (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Artery dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral arterial stenosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Iliac artery embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Total (Renal and urinary disorders) | 22 (22) | 27 (27) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 16 (16) | 18 (18) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 5 (5) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 3 (3) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Total (Gastrointestinal disorders) | 7 (7) | 15 (16) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Total (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 13 (13) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Total (Blood and lymphatic system disorders) | 5 (5) | 12 (12) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Total (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 8 (8) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
T-cell prolymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Total (Investigations) | 6 (6) | 7 (7) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 3 (3) | 0 (0)
Electrocardiogram PR prolongation (Investigations) | 2 (2) | 2 (2) | 0 (0)
Echocardiogram abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0)
Total (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Marasmus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Total (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatorenal failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Total (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Total (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lotus Valve (30 Day Follow Up) (N=1014) | Lotus Valve (1 Year Follow Up) (N=1014) | Lotus With Depth Guard (30 Day Follow Up) (N=50)
Bundle branch block left (Cardiac disorders) | 85 (86) | 88 (89) | 4 (4)
Catheter site haematoma (General disorders) | 11 (11) | 11 (11) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT02031302/Prot_SAP_000.pdf